CLINICAL TRIAL: NCT01794845
Title: Phase II Trial Using Erbitux+ Taxotere With Low Dose Fractionated Radiation for Recurrent Unresectable Locally Advanced Head and Neck Carcinoma
Brief Title: Cetuximab + Taxotere With Low Dose Fractionated Radiation for Head and Neck Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to lack of efficacy (overall response)
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Matthew Abramowitz, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090467
Record Dates: First submitted 2013-02-14; First posted 2013-02-20 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Squamous Cell Carcinoma; Head and Neck Cancer; Recurrent Disease
Keywords: SCCHN; Head and Neck Cancer; Squamous Cell Carcinoma; Recurrent
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Recurrence | interventions — Cetuximab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erbitux, Taxotere, LD Fractionated RT (Experimental): Erbitux, Taxotere and Low Dose Fractionated Radiation Therapy (LDFRT)
  Interventions: Drug: Erbitux; Drug: Taxotere; Radiation: Low Dose Fractionated Radiation Therapy

INTERVENTIONS:
Drug: Erbitux — Erbitux: 400 mg/m2 as a loading dose one week prior to radiation and taxotere, and then at 250 mg/m2 given weekly on Day 1 of treatment week following Taxotere.
  Other Names: Cetuximab
Drug: Taxotere — Taxotere : 20 mg/m2 IV once a week on Day 1 during treatment weeks 2 to 7.
  Other Names: Docetaxel
Radiation: Low Dose Fractionated Radiation Therapy — Low-dose fractionated Radiation (LDFRT): 0.5 Gy per fraction twice-a-day (BID) at least 6 to 8 hours apart on Days 2 and 3 of treatment weeks 2 to 7 for a total dose of 12 Gy.
  Other Names: LDFRT

SUMMARY:
Whether low-dose radiation in addition to Taxotere and Erbitux improves the response rate of patients with recurrent unresectable head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
The investigator's approach is based on the following reasons:

* Low dose hyper-radiation sensitivity response will be significantly enhanced in Taxotere- induced G2/M cell cycle arrest.
* LDFRT will render enhanced bax activation mediated mode of cell death.
* Erbitux will arrest the cells in G1/G0 phase leading to p21-mediated mode of cell death.
* The toxicity profile is expected to be minimal.

Based on the above mentioned reasons, we propose this novel schema of treatment in recurrent SCCHN.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed recurrence (reappearance of previously cleared) squamous cell cancer primary in the upper aerodigestive tract .Patients may have experienced more than one recurrence as long as the first recurrence occurred ≥ 6 months following the end of the prior RT.
2. The recurrence must have defined bi- or uni-dimensional measurements.
3. Recurrence must be confined to the head and neck above the clavicles (loco-regional recurrence).
4. The patient must not be a candidate for surgical resection.
5. Patients must be at least 6 months from completion of prior chemotherapy and radiation therapy.
6. Patients may have received prior chemotherapy as a component of their primary treatment, but not for recurrent disease.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
8. Granulocytes ≥ 1500/mm3, platelets ≥ 100,000/mm3, serum bilirubin ≤ 1.5 mg/dl, creatinine < 1.5 mg/dl within 3 weeks prior to registration.
9. Liver Function Tests (LFTs) ≤ 2 x normal (serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic-pyruvic transaminase (SGPT)/Alkaline Phosphatase). If > 2 x normal, liver ultrasound or CT is required to exclude metastases. If negative for metastases, patients are eligible.
10. Patients must sign a study-specific informed consent form prior to study entry.

Exclusion Criteria:

1. Distant metastases outside of the head and neck.
2. Primary disease in the nasopharynx or the salivary gland.
3. Other concurrent invasive malignancies.
4. Prior invasive malignancy unless disease free for at least two years (except prior in situ malignancies, e.g. cervix, breast, non-melanomatous skin cancer, etc. are permissible).
5. Intercurrent medical illnesses which would impair patient tolerance to therapy or limit survival.
6. Pre-existing grade ≥ 2 peripheral sensory neuropathy
7. Pregnant and nursing women are excluded because of the potential teratogenic effects and potential unknown effects on nursing newborns.
8. Prior history of sever hypersensitivity reaction to Docetaxol, Cetuximab or a drug with formulated with Polysorbate 80.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Abramowitz, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Erbitux, Taxotere, LD Fractionated RT: Erbitux, Taxotere and Low Dose Fractionated Radiation Therapy (LDFRT):
  * Erbitux: 400 mg/m2 as a loading dose one week prior to radiation and taxotere, and then at 250 mg/m2 given weekly on Day 1 of treatment week following Taxotere.
  * Taxotere: 20 mg/m2 IV once a week on Day 1 during treatment weeks 2 to 7.
  * Low-dose fractionated Radiation (LDFRT): 0.5 Gy per fraction twice-a-day (BID) at least 6 to 8 hours apart on Days 2 and 3 of treatment weeks 2 to 7 for a total dose of 12 Gy.
Period: Overall Study
Arm/Group | Erbitux, Taxotere, LD Fractionated RT
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erbitux, Taxotere, LD Fractionated RT
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants] — Population: Data for 4 of 5 participants analyzed due to 1 subject withdrawing prior to receiving protocol therapy.
  Participants
    number analyzed (Participants) | 4
    <=18 years | 0
    Between 18 and 65 years | 2
    >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data for 4 of 5 participants analyzed due to 1 subject withdrawing prior to receiving protocol therapy.
  Participants
    number analyzed (Participants) | 4
    Female | 0
    Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5
Site of Head and Neck Carcinoma [Count of Participants; unit: Participants] — Population: Data for 4 of 5 participants analyzed due to 1 subject withdrawing prior to receiving protocol therapy.
  Participants
    number analyzed (Participants) | 4
    Larynx | 2
    Floor of Mouth | 1
    Tonsil | 1
Surgery [Count of Participants; unit: Participants] — Number of study participants receiving surgery as treatment for primary tumor. Population: Data for 4 of 5 participants analyzed due to 1 subject withdrawing prior to receiving protocol therapy.
  Participants
    number analyzed (Participants) | 4
    (all) | 1
Chemotherapy [Count of Participants; unit: Participants] — Number of study participants receiving chemotherapy as treatment for primary tumor. Population: Data for 4 of 5 participants analyzed due to 1 subject withdrawing prior to receiving protocol therapy.
  Participants
    number analyzed (Participants) | 4
    (all) | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of Participants
Description: ORR is defined as the rate of study participants achieving complete response (CR) or partial response (PR) to protocol therapy according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) criteria.
Time Frame: Up to 6 months from End of Treatment, about 9 months
Population: Data for 4 of 5 participants analyzed due to 1 subject withdrawing prior to receiving protocol therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Erbitux, Taxotere, LD Fractionated RT
Number analyzed (Participants) | 4
percentage of participants
  Overall Response (CR+PR), 1 month | 50
  Overall Response (CR+PR), 6 months | 0
  Complete Response (CR), 1 month | 0
  Complete Response (CR), 6 months | 0
  Partial Response (PR), 1 month | 50
  Partial Response (PR), 6 months | 0
  Stable Disease (SD), 1 month | 25
  Stable Disease (SD), 6 months | 0
  Progressive Disease (PD), 1 month | 25
  Progressive Disease (PD), 6 months | 100

2. Secondary Outcome: Number of Study Participants Experiencing Treatment-Related Toxicity
Description: Assess the safety profile (acute and late toxicities) of the proposed treatment. Number of study participants experiencing treatment-related acute and late toxicity:
  * Acute toxicity is defined as toxicity occurring within 90 days of start of therapy.
  * Late/Long-term toxicity defined as toxicity occurring more than 90 days after start of therapy.
Time Frame: Up to 6 years
Population: Data for 4 of 5 participants analyzed due to 1 subject withdrawing prior to receiving protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Erbitux, Taxotere, LD Fractionated RT
Number analyzed (Participants) | 4
Participants
  Acute Toxicities | 4
  Late Toxicities | 0

3. Secondary Outcome: Estimated Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) is defined of the length of time from the start date of treatment to the earliest documented occurrence of disease progression according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) criteria. In the absence of an event constituting failure, follow up time will be censored at the date of last disease assessment.
Time Frame: Up to 6 years
Population: At the time of study termination in June 2016, 1 patient had already died, 1 patient had refused follow-up, 1 patient was lost to follow-up and 1 patient was alive with disease. Progression-free survival data were not analyzed due to an insufficient number of evaluable participants accrued and early study termination for lack of efficacy.
Arm/Group | Erbitux, Taxotere, LD Fractionated RT
Number analyzed (Participants) | 0

4. Secondary Outcome: Estimated Overall Survival (OS)
Description: Overall survival (OS) is defined as the length of time from the start of treatment that study participants diagnosed with the disease are still alive. OS will be measured from the start date of treatment to the date of death or last contact (censored observations).
Time Frame: Up to 6 years
Population: At the time of study termination in June 2016, 1 patient had already died, 1 patient had refused follow-up, 1 patient was lost to follow-up and 1 patient was alive with disease. Overall survival data were not analyzed due to an insufficient number of evaluable participants accrued and early study termination for lack of efficacy.
Arm/Group | Erbitux, Taxotere, LD Fractionated RT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Erbitux, Taxotere, LD Fractionated RT
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erbitux, Taxotere, LD Fractionated RT (N=4)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erbitux, Taxotere, LD Fractionated RT (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Pain (General disorders) | 1 (2)
Paronychia (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (7)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Data analyzed for 4 out of 5 study participants due to 1 study participant withdrawing prior to receiving study therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes